CLINICAL TRIAL: NCT04298567
Title: A Phase IV Study to Investigate the Safety and Effectiveness of Rivaroxaban(Xarelto) 2.5mg [BID]+Acetylsalicylic Acid(ASA) 75mg [OD] in Indian Patients With Coronary and/or Symptomatic Peripheral Artery Disease
Brief Title: Study to Learn More About the Safety and Effectiveness of Rivaroxaban (Xarelto) When Given Together With Acetylsalicylic Acid to Indian People With Narrowing of the Arteries of the Heart (CAD) and/or With Reduced Blood Flow in the Arteries of the Legs and Arms With Symptoms (Symptomatic PAD)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21269
Record Dates: First submitted 2020-02-19; First posted 2020-03-06 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Prevention of Atherothrombotic Events; Coronary Artery Disease (CAD); Symptomatic Peripheral Artery Disease (Symptomatic PAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Female and male patients with a diagnosis of CAD or symptomatic PAD will be enrolled within 4 weeks after the decision for treatment with rivaroxaban 2.5mg [BID] plus ASA 75mg [OD] has been made by the investigator.
  Interventions: Drug: Rivaroxaban (Xarelto,Bay 59-7939); Drug: Acetylsalicylic acid(ASA)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto,Bay 59-7939) — Rivaroxaban (2.5 mg [BID])
Drug: Acetylsalicylic acid(ASA) — ASA (75mg [QD]; dose according to local label.

SUMMARY:
This is an observational study in which data from Indian people with coronary artery disease and / or symptomatic peripheral artery disease who will be receiving the drug rivaroxaban (Xarelto) are studied.

Coronary artery disease (CAD) is a condition where the arteries that bring blood and oxygen to the heart become hardened and narrow. Peripheral artery disease (PAD) is a condition with reduced blood flow in the arteries of the legs and arms. People with CAD and / or PAD with symptoms may receive rivaroxaban from their doctors to prevent problems (for example, stoke) caused by blood clots and hardening of the arteries.

In this study researcher want to gather more information on the safety and the effectiveness of rivaroxaban when given together with the drug acetylsalicylic acid (also known as "aspirin") to people with CAD and / or PAD with symptoms in the routine practice in India. Researchers are especially interested whether patients under treatment experience any events such as minor or major bleedings, stroke, sickness of the heart or blood vessels. In addition, information on why and when treating doctors decide to start or stop the treatment with rivaroxaban and acetylsalicylic acid is of interest to the researchers.

The study plans to enroll about 300 male or female patients who are at least 18 years old and are already treated with the two drugs or at least with rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patient.
* Diagnosis of CAD or PAD.
* Treatment with Rivaroxaban 2.5mg tablet, co administered with acetylsalicylic acid (ASA), for the prevention of atherothrombotic events in adult patients with coronary artery disease (CAD) or symptomatic peripheral artery disease (PAD) at high risk of ischaemic events within 4 weeks prior to enrolment. also patients already on rivaroxaban treatment for ACS, who are subsequently fulfilling criteria for CAD, are allowed to be enrolled within 4 weeks of this decision being made.
* Patients who are willing to participate in this study (signed informed consent).

Exclusion Criteria:

* Contra-indications according to the local marketing authorization.
* Patients who will be treated with chronic anticoagulation therapy other than rivaroxaban 2.5mg given for CAD/PAD.
* Participation in an interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients with a diagnosis of CAD or symptomatic PAD will be enrolled within 4 weeks after the decision for treatment with rivaroxaban plus ASA has been made by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with haemorrhagic events and complications | Up to 13 months
  Consisting of minor and major bleeding events. The major bleeding complications are collected according to the International Society on Thrombosis and Haemostasis (ISTH) criteria as a composite of fatal bleeding, symptomatic bleeding into a critical organ (such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome), bleeding into surgical site requiring reoperation, bleeding leading to hospitalization.

SECONDARY OUTCOMES:
Number of participants with major adverse cardiovascular events (MACE) | Up to 13 months
  MACE: composite of MI, stroke, and cardiovascular death (and single components)
Number of participants with major adverse limb events (MALE) | Up to 13 months
  MALE: Major adverse limb events, incl. major amputation (and single components), and antithrombotic treatment patterns after MALE
Number of participants with thromboembolic events | Up to 13 months
  Thromboembolic events includes systemic embolism, venous thromboembolism
Number of participants with cardiovascular mortality | Up to 13 months
Number of participants with all-cause mortality | Up to 13 months
Number of participants with cardiac revascularization procedures | Up to 13 months
  Cardiac revascularization procedure includes Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Grafting (CABG)
Number of participants with peripheral revascularization procedures | Up to 13 months
Number of participants with carotid revascularization procedures | Up to 13 months
Duration of hospitalizations | Up to 13 months
  Hospitalizations includes stroke, cardiovascular reasons, MALE, or bleeding complications.
Total and pain free walking distance per individual for PAD patients | Change from baseline up to 13 months
Number of participants with history and diagnosis of CAD or PAD | Up to 13 months
  History and diagnosis of CAD, incl. history of myocardial infarction and vessel status.
  History and diagnosis of PAD, incl. ankle-brachial index (ABI).
Number of participants with individual risk | Up to 13 months
  Individual Risk classification: Co-morbidities (e.g. worsening symptoms, diabetes mellitus, chronic heart failure (CHF) renal impairment (eGFR <60 ml/min), Cerebrovascular disease(, ≥ 2 peripheral vascular beds affected, intermittent claudication, ABI <0.9, smoking, hypertension, hyperlipidaemia, carotid stenosis), and routinely collected key laboratory data.
Number of participants with revascularization procedures and prior interventions (PCI, CABG), peripheral revascularization procedures | Up to 13 months
Type of prior and concomitant antithrombotic treatment and other secondary prevention therapies in patients with CAD or PAD | Up to 13 months
Dose of prior and concomitant antithrombotic treatment and other secondary prevention therapies in patients with CAD or PAD | Up to 13 months
Duration of prior and concomitant antithrombotic treatment and other secondary prevention therapies in patients with CAD or PAD | Up to 13 months
Reasons and decision points for introducing rivaroxaban 2.5 mg [BID] | Up to 13 months
  BID: twice per day dosing
Reasons for discontinuation of rivaroxaban 2.5 mg [BID]. | Up to 13 months
Planned and actual duration of treatment with rivaroxaban 2.5 mg [BID]. | Up to 13 months
Planned and actual duration of treatment with ASA 75 mg [OD] | Up to 13 months
  QD:once per day dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.